CLINICAL TRIAL: NCT02133131
Title: A Phase II Open-Label Clinical Trial to Study the Efficacy and Safety of the Combination Regimen of MK-5172, MK-8742, and Sofosbuvir in Treatment-Naïve Subjects With Chronic HCV GT1 or GT3 Infection
Brief Title: Efficacy and Safety of Grazoprevir (MK-5172), Elbasvir (MK-8742), and Sofosbuvir for Chronic Infection With Hepatitis C Virus Genotypes 1 and 3 (MK-5172-074)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5172-074
Record Dates: First submitted 2014-05-05; First posted 2014-05-07 (Estimated); Results first posted 2016-11-17 (Estimated); Last update posted 2021-02-05 (Actual); Status verified 2021-01

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — grazoprevir; elbasvir-grazoprevir drug combination; Sofosbuvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (7):
- GT1:NC Grazoprevir/Elbasvir+SOF 4wk (Experimental): Participants took grazoprevir/elbasvir (100mg/50mg) FDC with SOF 400mg once daily (q.d.) by mouth for 4 weeks (n=30 planned).
  Interventions: Drug: Grazoprevir/Elbasvir FDC; Drug: Sofosbuvir
- GT1:NC Grazoprevir/Elbasvir+SOF 6wk (Experimental): Participants took grazoprevir/elbasvir (100mg/50mg) FDC + SOF 400mg q.d. by mouth for 6 weeks (n=30 planned).
  Interventions: Drug: Grazoprevir/Elbasvir FDC; Drug: Sofosbuvir
- GT1:C Grazoprevir/Elbasvir+SOF 6wk (Experimental): Participants took grazoprevir/elbasvir (100mg/50mg) FDC + SOF 400mg q.d. by mouth for 6 weeks (n=20 planned).
  Interventions: Drug: Grazoprevir/Elbasvir FDC; Drug: Sofosbuvir
- GT1:C Grazoprevir/Elbasvir+SOF 8wk (Experimental): Participants took grazoprevir/elbasvir (100mg/50mg) FDC + SOF 400mg q.d. by mouth for 8 weeks (n=20 planned).
  Interventions: Drug: Grazoprevir/Elbasvir FDC; Drug: Sofosbuvir
- GT3:NC Grazoprevir/Elbasvir+SOF 8wk (Experimental): Participants took grazoprevir/elbasvir (100mg/50mg) FDC + SOF 400mg q.d. by mouth for 8 weeks (n=15 planned).
  Interventions: Drug: Grazoprevir/Elbasvir FDC; Drug: Sofosbuvir
- GT3:NC Grazoprevir/Elbasvir+SOF 12wk (Experimental): Participants took grazoprevir/elbasvir (100mg/50mg) FDC + SOF 400mg q.d. by mouth for 12 weeks (n=15 planned).
  Interventions: Drug: Grazoprevir/Elbasvir FDC; Drug: Sofosbuvir
- GT3:C Grazoprevir/Elbasvir+SOF 12wk (Experimental): Participants took grazoprevir/elbasvir (100mg/50mg) FDC + SOF 400mg q.d. by mouth for 12 weeks (n=10 planned).
  Interventions: Drug: Grazoprevir/Elbasvir FDC; Drug: Sofosbuvir

INTERVENTIONS:
Drug: Grazoprevir/Elbasvir FDC — FDC tablet containing grazoprevir 100 mg + elbasvir 50 mg taken q.d. by mouth.
  Other Names: MK-5172A, Zepatier
Drug: Sofosbuvir — Sofosbuvir 400mg tablet taken q.d. by mouth.

SUMMARY:
This is a study of grazoprevir (MK-5172) + elbasvir (MK-8742) and sofosbuvir (SOF) in treatment-naive participants with chronic hepatitis C (HCV) genotype (GT) 1 or GT3. The objective is to determine the proportion of participants achieving sustained virologic response 12 weeks after ending study treatment (SVR12).

DETAILED DESCRIPTION:
The study is an open-label, single-center, multiple-arm investigation of a fixed-dose combination [FDC] of grazoprevir 100mg + elbasvir 50mg, and SOF 400mg, in treatment-naive participants with chronic HCV GT1 or GT3. The impact of study treatment regimens of varying duration on SVR12 (undetectable HCV ribonucleic acid [RNA] 12 weeks after ending study treatment) in cirrhotic (C) participants and non-cirrhotic (NC) participants will be determined (Part A). Any HCV GT1 participant from study Arms 1-4 in Part A who experienced virologic relapse will be offered retreatment consisting of 12 additional weeks of treatment with MK-5172/MK-8742 + SOF + ribavirin and 24 weeks of follow-up in Part B.

ELIGIBILITY:
Inclusion Criteria:

* has HCV RNA ≥10,000 IU/mL in peripheral blood at the time of screening
* has documented chronic HCV GT1 or GT3 infection
* has either negative or positive history of liver cirrhosis based on liver biopsy, Fibroscan, or FibroSure ® (Fibrotest®)
* is treatment naïve to all anti-HCV treatment

Exclusion Criteria:

* has evidence of decompensated liver disease
* is coinfected with hepatitis B virus (e.g. hepatitis B surface antigen positive) or human immunodeficiency virus
* has a history of malignancy ≤5 years prior to signing informed consent, or is under evaluation for other active or suspected malignancy
* has cirrhosis and liver imaging within 6 months of Day 1 showing evidence of hepatocellular carcinoma (HCC) or is under evaluation for HCC
* has clinically-relevant drug or alcohol abuse within 12 months of screening
* has any of the following conditions: organ transplants other than cornea and hair, poor venous access that precludes routine peripheral blood sampling, history of gastric surgery or malabsorption disorders, or any medical condition requiring, or likely to require, chronic systemic administration of corticosteroids during the course of the trial
* has a history of chronic hepatitis not caused by HCV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2014-06-13 (Actual); Primary Completion 2015-11-02 (Actual); Study Completion 2016-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Lawitz E, Poordad F, Gutierrez JA, Wells JT, Landaverde CE, Evans B, Howe A, Huang HC, Li JJ, Hwang P, Dutko FJ, Robertson M, Wahl J, Barr E, Haber B. Short-duration treatment with elbasvir/grazoprevir and sofosbuvir for hepatitis C: A randomized trial. Hepatology. 2017 Feb;65(2):439-450. doi: 10.1002/hep.28877. Epub 2016 Dec 19. PMID 27770561

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The current interim disclosure covers data up to 12 weeks after completing study treatment. The cutoff date for this initial disclosure is 12-Feb-2015. GT3 participants have completed treatment but are ongoing in follow-up.
Groups:
- GT1: NC Grazoprevir/Elbasvir + SOF 4 Weeks: HCV GT1 NC participants took grazoprevir 100 mg + elbasvir 50 mg FDC with SOF 400 mg for 4 weeks.
- GT1: NC Grazoprevir/Elbasvir + SOF 6 Weeks: HCV GT1 NC participants took grazoprevir 100 mg + elbasvir 50 mg FDC with SOF 400 mg for 6 weeks.
- GT1: C Grazoprevir/Elbasvir + SOF 6 Weeks: HCV GT1 C participants took grazoprevir 100 mg + elbasvir 50 mg FDC with SOF 400 mg for 6 weeks.
- GT1: C Grazoprevir/Elbasvir + SOF 8 Weeks: HCV GT1 C participants took grazoprevir 100 mg + elbasvir 50 mg FDC with SOF 400 mg for 8 weeks.
- GT3: NC Grazoprevir/Elbasvir + SOF 8 Weeks: HCV GT3 NC participants took grazoprevir 100 mg + elbasvir 50 mg FDC with SOF 400 mg for 8 weeks.
- GT3: NC Grazoprevir/Elbasvir + SOF 12 Weeks: HCV GT3 NC participants took grazoprevir 100 mg + elbasvir 50 mg FDC with SOF 400 mg for 12 weeks.
- GT3: C Grazoprevir/Elbasvir + SOF 12 Weeks: HCV GT3 C participants took grazoprevir 100 mg + elbasvir 50 mg FDC with SOF 400 mg for 12 weeks.
Period: Overall Study
Arm/Group | GT1: NC Grazoprevir/Elbasvir + SOF 4 Weeks | GT1: NC Grazoprevir/Elbasvir + SOF 6 Weeks | GT1: C Grazoprevir/Elbasvir + SOF 6 Weeks | GT1: C Grazoprevir/Elbasvir + SOF 8 Weeks | GT3: NC Grazoprevir/Elbasvir + SOF 8 Weeks | GT3: NC Grazoprevir/Elbasvir + SOF 12 Weeks | GT3: C Grazoprevir/Elbasvir + SOF 12 Weeks
Started | 31 | 30 | 20 | 21 | 15 | 14 | 12
Completed | 26 | 25 | 19 | 15 | 0 | 0 | 0
Not Completed | 5 | 5 | 1 | 6 | 15 | 14 | 12
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Status not recorded | 4 | 5 | 1 | 4 | 0 | 0 | 0
Not completed — Ongoing in study | 0 | 0 | 0 | 0 | 15 | 14 | 11
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GT1: NC Grazoprevir/Elbasvir + SOF 4 Weeks | GT1: NC Grazoprevir/Elbasvir + SOF 6 Weeks | GT1: C Grazoprevir/Elbasvir + SOF 6 Weeks | GT1: C Grazoprevir/Elbasvir + SOF 8 Weeks | GT3: NC Grazoprevir/Elbasvir + SOF 8 Weeks | GT3: NC Grazoprevir/Elbasvir + SOF 12 Weeks | GT3: C Grazoprevir/Elbasvir + SOF 12 Weeks | Total
Number analyzed (Participants) | 31 | 30 | 20 | 21 | 15 | 14 | 12 | 143
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.1 (9.7) | 51.2 (9.5) | 55.7 (7.7) | 56.8 (8.8) | 51.3 (10.1) | 42.2 (11.7) | 55.3 (5.3) | 52.3 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 7 | 8 | 4 | 6 | 2 | 49
  Male | 20 | 19 | 13 | 13 | 11 | 8 | 10 | 94

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Viral Response (SVR) 12 Weeks After Completing All Study Therapy (SVR12)
Description: The percentage of participants achieving SVR12, defined as HCV ribonucleic acid (RNA) <15 IU/mL 12 weeks after completing all study therapy, was determined for each arm. Plasma levels of HCV RNA were measured using the Roche COBAS© AmpliPrep/COBAS© TaqMan© HCV Test v. 2.0.
Time Frame: Up to 24 weeks
Population: The Per Protocol (PP) population includes all randomized and treated participants who did not have protocol deviations that may substantially affect the results of the primary and secondary endpoints.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | GT1: NC Grazoprevir/Elbasvir + SOF 4 Weeks | GT1: NC Grazoprevir/Elbasvir + SOF 6 Weeks | GT1: C Grazoprevir/Elbasvir + SOF 6 Weeks | GT1: C Grazoprevir/Elbasvir + SOF 8 Weeks | GT3: NC Grazoprevir/Elbasvir + SOF 8 Weeks | GT3: NC Grazoprevir/Elbasvir + SOF 12 Weeks | GT3: C Grazoprevir/Elbasvir + SOF 12 Weeks
Number analyzed (Participants) | 30 | 28 | 20 | 19 | 15 | 14 | 11
Percentage of participants | 33.3 [17.3 to 52.8] | 89.3 [71.8 to 97.7] | 80.0 [56.3 to 94.3] | 89.5 [66.9 to 98.7] | 93.3 [68.1 to 99.8] | 100.0 [76.8 to 100.00] | 90.9 [58.7 to 99.8]

2. Primary Outcome: Number of Participants Experiencing at Least 1 Adverse Event (AE)
Description: An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment.
Time Frame: Up to Week 14
Population: The All Participants as Treated (APaT) population consists of all participants who received ≥1 dose of study drug.
Measure: Number; unit: Number of participants
Arm/Group | GT1: NC Grazoprevir/Elbasvir + SOF 4 Weeks | GT1: NC Grazoprevir/Elbasvir + SOF 6 Weeks | GT1: C Grazoprevir/Elbasvir + SOF 6 Weeks | GT1: C Grazoprevir/Elbasvir + SOF 8 Weeks | GT3: NC Grazoprevir/Elbasvir + SOF 8 Weeks | GT3: NC Grazoprevir/Elbasvir + SOF 12 Weeks | GT3: C Grazoprevir/Elbasvir + SOF 12 Weeks
Number analyzed (Participants) | 31 | 30 | 20 | 21 | 15 | 14 | 12
Number of participants | 5 | 7 | 7 | 4 | 4 | 3 | 3

3. Primary Outcome: Number of Participants Discontinuing Study Therapy Due to an AE
Description: as for outcome 2
Time Frame: Up to Week 12
Population: The APaT population consists of all participants who received ≥1 dose of study drug.
Measure: Number; unit: Number of participants
Arm/Group | GT1: NC Grazoprevir/Elbasvir + SOF 4 Weeks | GT1: NC Grazoprevir/Elbasvir + SOF 6 Weeks | GT1: C Grazoprevir/Elbasvir + SOF 6 Weeks | GT1: C Grazoprevir/Elbasvir + SOF 8 Weeks | GT3: NC Grazoprevir/Elbasvir + SOF 8 Weeks | GT3: NC Grazoprevir/Elbasvir + SOF 12 Weeks | GT3: C Grazoprevir/Elbasvir + SOF 12 Weeks
Number analyzed (Participants) | 31 | 30 | 20 | 21 | 15 | 14 | 12
Number of participants | 0 | 0 | 0 | 1 | 0 | 0 | 0

4. Secondary Outcome: Percentage of Participants Achieving SVR 4 Weeks After Completing All Study Therapy (SVR4)
Description: The percentage of participants achieving SVR4, defined as HCV ribonucleic acid (RNA) <15 IU/mL 4 weeks after completing all study therapy, was determined for each arm. Plasma levels of HCV RNA were measured using the Roche COBAS© AmpliPrep/COBAS© TaqMan© HCV Test v. 2.0.
Time Frame: Up to 16 weeks
Population: Analysis of SVR4 is ongoing and results will be indicated in a future report.
Arm/Group | GT1: NC Grazoprevir/Elbasvir + SOF 4 Weeks | GT1: NC Grazoprevir/Elbasvir + SOF 6 Weeks | GT1: C Grazoprevir/Elbasvir + SOF 6 Weeks | GT1: C Grazoprevir/Elbasvir + SOF 8 Weeks | GT3: NC Grazoprevir/Elbasvir + SOF 8 Weeks | GT3: NC Grazoprevir/Elbasvir + SOF 12 Weeks | GT3: C Grazoprevir/Elbasvir + SOF 12 Weeks
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 14 weeks
Description: An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment.
Arm/Group | GT1: NC Grazoprevir/Elbasvir + SOF 4 Weeks | GT1: NC Grazoprevir/Elbasvir + SOF 6 Weeks | GT1: C Grazoprevir/Elbasvir + SOF 6 Weeks | GT1: C Grazoprevir/Elbasvir + SOF 8 Weeks | GT3: NC Grazoprevir/Elbasvir + SOF 8 Weeks | GT3: NC Grazoprevir/Elbasvir + SOF 12 Weeks | GT3: C Grazoprevir/Elbasvir + SOF 12 Weeks
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/30 | 1/20 | 1/21 | 1/15 | 0/14 | 1/12
Other Adverse Events (participants affected / at risk) | 2/31 | 2/30 | 2/20 | 4/21 | 4/15 | 3/14 | 3/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GT1: NC Grazoprevir/Elbasvir + SOF 4 Weeks (N=31) | GT1: NC Grazoprevir/Elbasvir + SOF 6 Weeks (N=30) | GT1: C Grazoprevir/Elbasvir + SOF 6 Weeks (N=20) | GT1: C Grazoprevir/Elbasvir + SOF 8 Weeks (N=21) | GT3: NC Grazoprevir/Elbasvir + SOF 8 Weeks (N=15) | GT3: NC Grazoprevir/Elbasvir + SOF 12 Weeks (N=14) | GT3: C Grazoprevir/Elbasvir + SOF 12 Weeks (N=12)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic mass (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lobar pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GT1: NC Grazoprevir/Elbasvir + SOF 4 Weeks (N=31) | GT1: NC Grazoprevir/Elbasvir + SOF 6 Weeks (N=30) | GT1: C Grazoprevir/Elbasvir + SOF 6 Weeks (N=20) | GT1: C Grazoprevir/Elbasvir + SOF 8 Weeks (N=21) | GT3: NC Grazoprevir/Elbasvir + SOF 8 Weeks (N=15) | GT3: NC Grazoprevir/Elbasvir + SOF 12 Weeks (N=14) | GT3: C Grazoprevir/Elbasvir + SOF 12 Weeks (N=12)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Fatigue (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation.